CLINICAL TRIAL: NCT06295601
Title: Effect of Telerehabilitation-Based Motor Imagery and Action Observation Training on Balance and Functional Mobility in Multiple Sclerosis: Randomized Controlled Study
Brief Title: Telerehabilitation Based Motor Imagery and Action Observation Training in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/5591
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: motor imagery; telerehabilitation; action observation therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Individuals will receive standard rehabilitation and telerehabilitation-based motor imagery and action observation therapy.
  Interventions: Other: Traditional rehabilitation; Other: Action observation therapy and motor imagery
- Control group (Experimental): Individuals will receive standard rehabilitation.
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Other: Traditional rehabilitation — The program consists of a joint treatment in which lower extremity strengthening and balance exercises are carried out synchronously. The program will include a total of 5 minutes of warm-up, 5 minutes of cool-down and 30 minutes of exercises related to the program. The difficulty of the program will increase by changing the number of exercises and increasing the weight in strengthening exercises. Progress in balance and coordination exercises will vary by changing the ground, increasing the standing time, and keeping the eyes open and closed.
Other: Action observation therapy and motor imagery — In the experimental group, in addition to traditional telerehabilitation, action observation and motor imagery of 4 exercises will be performed in each session. A video will be prepared for 4 exercises. Then, the participant will perform 2 minutes of action observation of each movement, followed by 1 minute of motor imagery. In addition to the traditional telerehabilitation program, a 12-minute combination of action observation and motor imagery will be performed in each session. Exercises will be changed every two weeks, gradually increasing the difficulty.
  Arms: Experimental group

SUMMARY:
This study aims to investigate the effects of the treatment combination consisting of motor imagery and action observation therapy on balance, functional mobility, lower extremity muscle strength, fatigue and quality of life.

DETAILED DESCRIPTION:
The study population was participants with relapsing remitting multiple sclerosis. The traditional rehabilitation program consists of a joint treatment in which lower extremity strengthening and balance exercises are carried out synchronously for the experimental and control groups. Motor imagery and action observation therapy based on telerehabilitation of certain movements will be applied to the experimental group. All treatments will be carried out online via the zoom program. The treatment program will be applied 3 times a week for 6 weeks. Evaluations will be made before and after the treatment program. Assessments include balance, lower extremity muscle strength and functional mobility, fatigue, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mulltiple sclerosis according to the McDonald criteria
* Expanded Disability Status Scale<5.5,
* Being between the ages of 18-65,
* Mini mental test score>24,
* Have a phone that can adapt to participating in a video call

Exclusion Criteria:

* Having another additional neurological disease that may cause balance and coordination disorders,
* Receiving physical therapy in the last 6 months,
* Having an attack in the last 3 months
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline
  Berg Balance Scale consists of a total of 14 items. Evaluation for each stage is made between 0-4. Higher score indicates better functional balance performance
Berg Balance Scale | 6 weeks after baseline
  Berg Balance Scale consists of a total of 14 items. Evaluation for each stage is made between 0-4. Higher score indicates better functional balance performance
Muscle strength and functional mobility | Baseline
  The participant will be asked to sit and stand up from a standard chair between 42-45 cm, with hands crossed on the chest, without support, 5 times. The time will be stopped when the participant completes the last sitting. It will be recorded in seconds.
Muscle strength and functional mobility | 6 weeks after baseline
  The participant will be asked to sit and stand up from a standard chair between 42-45 cm, with hands crossed on the chest, without support, 5 times. The time will be stopped when the participant completes the last sitting. It will be recorded in seconds.

SECONDARY OUTCOMES:
Fatigue Severity Scale | Baseline
  This scale consists of a total of 9 items and is scored between 0-7. >4 points indicate fatigue
Fatigue Severity Scale | 6 weeks after baseline
  This scale consists of a total of 9 items and is scored between 0-7. >4 points indicate fatigue
Multiple Sclerosis International Quality of Life (MusiQoL) questionnaire | Baseline
  The scale consists of 31 questions in 9 dimensions (subscales). The index score is calculated as the average of these subscale scores. All 9 dimensions and the index score are linearly transformed and standardized on a scale from 0 to 100; where 0 indicates the worst possible level of quality of life and 100 indicates the best level.
Multiple Sclerosis International Quality of Life (MusiQoL) questionnaire | 6 weeks after baseline
  The scale consists of 31 questions in 9 dimensions (subscales). The index score is calculated as the average of these subscale scores. All 9 dimensions and the index score are linearly transformed and standardized on a scale from 0 to 100; where 0 indicates the worst possible level of quality of life and 100 indicates the best level.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu talu, Study Director — Inonu University

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared with other researchers if desired.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study was published
Access Criteria: If requested from the authors, it can be shared with researchers at the authors' discretion.